CLINICAL TRIAL: NCT06793800
Title: Effect of TAVNS Application on Respiratory Functions in Stroke Patients
Brief Title: Effect of Transcutaneous Auricular Vagus Nerve Stimulation Application on Respiratory Functions in Stroke Patients
Acronym: TAVNS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Burcu AKKURT, Assistant Professor, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 80.2024fbu
Record Dates: First submitted 2025-01-21; First posted 2025-01-27 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Hemiplegia; Respiratory Function Loss
Keywords: hemiplegia; Vagus Nerve Stimulation; Respiration
MeSH Terms: conditions — Hemiplegia; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: Two groups with experimental group (TAVSS + conventional physiotherapy) and sham TAVSS + (conventional physiotherapy)
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants will not be aware of which group they are assigned to. The treatment protocols, evaluations, and statistical calculations will be carried out by three separate investigators.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (TAVSS + conventional physiotherapy) (Experimental): TAVSS and conventional physiotherapy will be applied for a total of 10 sessions, three times a week. TAVSS application electrodes will be placed on the tragus and the inner and posterior surfaces of the concha in both the right and left outer ear. The stimulation will be delivered continuously for 20 minutes with a biphasic asymmetric waveform, a pulse duration of 300 microseconds, and a frequency of 25 hertz. Electrical stimulation will be increased in 0.1 mA increments until the perception threshold is reached. Individualized conventional physiotherapy protocols tailored to the specific needs of the patients in the experimental group will be administered by a physiotherapist for a total of 10 sessions, three times a week. The conventional physiotherapy interventions will generally include strengthening exercises, stretching exercises, proprioceptive neuromuscular facilitation, electrotherapy, balance exercises, fine motor exercises, active range of motion exercises (45 minutes).
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- control (sham TAVSS + conventional physiotherapy) (Sham Comparator): shamTAVSS and conventional physiotherapy will be applied for a total of 10 sessions, three times a week. TAVSS application electrodes will be placed on the tragus and the inner and posterior surfaces of the concha in both the right and left outer ear without any current. Individualized conventional physiotherapy protocols tailored to the specific needs of the patients in this group will be administered by a physiotherapist for a total of 10 sessions, three times a week. The conventional physiotherapy interventions will generally include strengthening exercises, stretching exercises, proprioceptive neuromuscular facilitation, electrotherapy, balance exercises, fine motor exercises, active range of motion exercises (45 minutes).
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — TAVSS is an application system that uses an electrical transcutaneous stimulation device placed on the concha or tragus of the ear. Functional Magnetic Resonance Imaging studies have shown that stimulation of these areas activates the ipsilateral nucleus tractus solitarius (NTS) via vagal projections to the brainstem and forebrain. Unlike cervical vagus nerve stimulation, TAVSS utilizes a physiological pathway to activate the NTS and the dorsal motor nucleus, which subsequently sends impulses bilaterally to the heart surface via efferent cervical vagus nerves. Therefore, this technique eliminates the possibility of directly and asymmetrically stimulating cardiac motor efferent fibers, which could lead to adverse cardiac events. TAVSS combines advantageous qualities such as being non-invasive, cost-effective, convenient, and efficient.

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Transcutaneous Auricular Vagus Nerve Stimulation (TAVSS) in improving respiratory muscle strength and function in chronic stroke patients. It aims to explore TAVSS as a potential complementary approach in enhancing rehabilitation outcomes for this population.

DETAILED DESCRIPTION:
Introduction Stroke is one of the leading causes of morbidity and long-term disability worldwide. Respiratory muscle weakness is a common complication in stroke patients, leading to respiratory dysfunction, increased aspiration risk, and higher mortality. Post-stroke, reduced vital capacity, maximum inspiratory and expiratory pressure, and low expiratory reserve volume significantly affect respiratory muscle function.

Objective This study aims to investigate the effects of Transcutaneous Auricular Vagus Nerve Stimulation (TAVSS) on respiratory parameters in chronic stroke patients.

Participants and Methods

The study included 50 chronic stroke patients in their 1st to 3rd year post-stroke, meeting specific motor levels in Brunnstrom Staging.

Participants were randomized equally into experimental (TAVSS + conventional physiotherapy) and control (sham TAVSS + conventional physiotherapy) groups.

Treatment Protocol

Experimental Group: TAVSS and conventional physiotherapy were applied three times per week for a total of 10 sessions. TAVSS was delivered for 20 minutes using a biphasic asymmetric waveform.

Control Group: Sham TAVSS (without current) and conventional physiotherapy were applied with the same frequency and duration.

Both groups received individualized physiotherapy protocols, including strengthening, stretching, balance exercises, electrotherapy, and neurodevelopmental treatment.

Measurements and Evaluation

Chest circumference measurements were taken at the axillary, epigastric, and subcostal regions during deep inspiration and expiration using a tape measure.

Respiratory function parameters (Maximum Inspiratory Pressure, Maximum Expiratory Pressure, Forced Expiratory Volume in 1 Second, Forced Vital Capacity, Forced Expiratory Volume in 1 Second to Forced Vital Capacity Ratio) were measured using the Minispir 2 spirometer before treatment and after the 10th session.

Conclusion and Recommendations The study aims to evaluate the impact of TAVSS on improving respiratory muscle strength and function, presenting an alternative approach in stroke rehabilitation. TAVSS is expected to support respiratory function and positively influence rehabilitation outcomes in stroke patients

ELIGIBILITY:
Inclusion Criteria:

* Being a chronic stroke patient with an ischemic or hemorrhagic stroke diagnosis made 1-3 years ago
* Having been diagnosed with stroke for the first time
* Ability to understand and follow simple verbal instructions
* Being between the ages of 40 and 80
* No conditions affecting perioral muscles, such as facial paralysis or swallowing disorders
* No visual, auditory, or communication problems
* No cardiopulmonary disorders
* No additional neurological, cardiovascular, orthopedic, or similar conditions causing balance problems
* Mini Mental State Examination (MMSE) score ≥24
* No surgical operations or Botox applications in the last 6 months
* Scoring 2 or below on the Modified Ashworth Scale

Exclusion Criteria:

* Presence of infection, ulcer, or scar on the auricle
* Metallic implants in the skull, hypersensitivity, injury, or inflammation inside the ear
* Chronic pulmonary and/or cardiac diseases
* Resting heart rate below 60 beats per minute
* Devices such as pacemakers or cochlear implants
* Uncontrolled hypertension
* Chronic obstructive pulmonary disease (COPD) or asthma unrelated to stroke
* History of surgical operation or Botox application within the last 6 months
* Presence of aphasia, apraxia, or neglect syndrome
* History of 2 or more strokes (SVO)
* Comorbid conditions affecting respiratory functions (e.g., Multiple Sclerosis, Parkinson's, spinal cord injury, contractures, deformities after fractures, active upper or lower respiratory infections, etc.)
* Lack of cooperation

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2025-08-26 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Inspiratory muscle strength | From enrollment to the end of treatment at 4 weeks
  Inspiratory muscle strength will be measured using the Minispir 2 spirometer by Medical International Research. This spirometer, classified as a Class II medical device (medium risk) by Health Canada, is a non-invasive tool for assessing respiratory function. It evaluates lung ventilation by measuring the air volume during inspiration and expiration. The device records inspiratory effort and lung capacity, helping determine respiratory muscle performance.
Expiratory muscle strength | From enrollment to the end of treatment at 4 weeks
  Expiratory muscle strength will be measured using the Minispir 2 spirometer by Medical International Research. This spirometer, classified as a Class II medical device (medium risk) by Health Canada, is a non-invasive tool for assessing respiratory function. It evaluates lung ventilation by measuring air volume during expiration, helping assess expiratory muscle performance and overall pulmonary function.
Forced Expiratory Volume in 1 Second (FEV₁) | From enrollment to the end of treatment at 4 weeks
  Forced Expiratory Volume in 1 Second (FEV₁) will be measured using the Minispir 2 spirometer by Medical International Research. This spirometer, classified as a Class II medical device (medium risk) by Health Canada, is a non-invasive tool for assessing respiratory function. It evaluates lung ventilation by measuring the air volume exhaled in the first second of a forced expiration, providing critical data on airway obstruction and pulmonary function.
Forced Vital Capacity (FVC) | From enrollment to the end of treatment at 4 weeks
  Forced Vital Capacity (FVC) will be measured using the Minispir 2 spirometer by Medical International Research. This spirometer, classified as a Class II medical device (medium risk) by Health Canada, is a non-invasive tool for assessing respiratory function. It evaluates lung ventilation by measuring the maximum air volume forcefully exhaled after a deep inhalation, providing essential data on pulmonary function and lung capacity.
Forced Expiratory Volume in 1 Second (FEV₁) to Forced Vital Capacity (FVC) | From enrollment to the end of treatment at 4 weeks
  Forced Expiratory Volume in 1 Second (FEV₁) to Forced Vital Capacity (FVC) ratio will be measured using the Minispir 2 spirometer by Medical International Research. This spirometer, classified as a Class II medical device (medium risk) by Health Canada, is a non-invasive tool for assessing respiratory function. It evaluates lung ventilation by determining the proportion of air exhaled in the first second relative to total forced vital capacity, providing key insights into airway obstruction and pulmonary function.

SECONDARY OUTCOMES:
Chest Circumference Measurement | From enrollment to the end of treatment at 4 weeks
  The chest circumference of patients in the Experimental and Control groups will be measured during deep inspiration and expiration using a measuring tape. Measurements will be taken at the axillary, epigastric, and subcostal regions as both baseline (initial) and post-treatment (final) assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu AKKURT, Study Director — Fenerbahce University
Locations (1):
- Mediworld Medical Center Physical Therapy and Rehabilitation Department, Istanbul, Turkey (Türkiye)